CLINICAL TRIAL: NCT04551638
Title: Virtual-self Identity Construal in Online Video Games: A Repertory Grid Study
Status: Completed | Type: Observational
Sponsor: University of Barcelona (Other)
Collaborators: Universitat Oberta de Catalunya (Other)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, Professor, University of Barcelona
Other Study IDs: UBipcsagp
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: General Population
Keywords: Personal constructs; Immersion; Ideal self; Actual self; Virtual self; Avatar; Videogames; MMORPG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Online Videogame Players: One cohort of healthy young adults players of online video games.
  Interventions: Other: Psychological assessment with the Repertory Grid Technique

INTERVENTIONS:
Other: Psychological assessment with the Repertory Grid Technique — The RGT is a constructivist psychological tool to explore the structure and content of personal identity.
  Other Names: RGT

SUMMARY:
New technologies are changing the way of approach for many concepts that used to be quite established in the past. The Internet, and especially online videogames where people can create a customizable character to serve as their avatar on a virtual environment, seems to have a great impact on the way people construe their identity. People may use online gaming as a means to experience an enhanced version of their self that matches more accurately the attributes and traits they often relate to their ideal self or even other alternative selves.

With this project, the researchers aim to study the role that new technologies have on the way people build their identity nowadays. More specifically, the researchers intend to study how people use videogame avatars as a means to explore different alternative identities. The rebelieve that, it is possible for people to manifest entirely different versions of themselves through their online videogame characters. Sometimes, those alternative identities may even be a projection of what the player considers to be an ideal version of themselves. Other variables may increase or hinder that capacity to project the ideal self on a customizable "virtual self"; some are inherent to the person, such as cognitive complexity, their current level of psychological distress or their main motivation for playing, while others may be more related to the specific game they play, such as the degree of immersion experienced while playing.

The researchers will use the repertory grid technique to explore online videogame players' personal construct systems and how an ideal version of themselves and their perceived self-image may help to understand their need to explore alternative identities through their videogame characters. They will also administrate other instruments to measure people's experienced immersion when playing the game, the aspects of it that are more appealing to them, and their degree of subjective psychological distress in order to assess how these variables, among others extracted from the repertory grid, may affect this identity exploration.

DETAILED DESCRIPTION:
INTRODUCTION

Since the appearance of online videogames, there has been a growing interest in how people behave socially on virtual media that grants people the possibility of adopting a whole new identity as a customized character. A previous study observed a tendency from players to create their videogame character so that it would resemble more their ideal selves than their actual ones, and actually reported their virtual avatar as having more desirable personality traits than their actual self. Additionally, in a more recent study, it was observed that the level of immersion during gameplay and a high discrepancy between the ideal and actual selves favored that people created their virtual characters as more similar to their ideal self. Thus, people who are already satisfied with their actual self may instead tend to create a virtual self that is entirely different from both their actual and ideal selves. The mere fact of exploring different identities has been shown to be rewarding by itself, without the need for the new identities to fulfill any perceived limitations.

However, none of these studies has been conducted using a constructivist framework. Theories based on that framework, such as the Personal Construct Theory (PCT), provide a tailored assessment for each individual's perception of the world and themselves instead of classifying them into pre-established dimensions that may, or may not, belong to their meaning system. Based on this theory, the Repertory Grid Technique allows the assessment of the degree to which people perceive themselves as similar or different from other people, and their representation of what they would like to be (i.e., "ideal self"). Moreover, in the videogame research field, the PCT also permits to explore gamers' construal of their virtual self, and whether it resembles more their ideal self, their actual self, or none. From the repertory grid, other measures can also be extracted that will help on this research, such as their self-ideal discrepancy, which represents the distance between the actual self and the ideal self, the presence of cognitive conflicts within participants' construct systems, or their interpersonal construct differentiation, defined as the tendency of a construct system to perceive the self and other elements through several dimensions, with different nuances (an indicator of cognitive complexity). For this project, the researchers will extract two additional measures as a result of including the virtual self in the participants' grid. These measures are the self-virtual discrepancy, understood as the distance between the actual self and the virtual self, and the virtual-ideal discrepancy, which is the distance between the virtual self and the ideal self. These measures will allow to assess to which degree the participants' videogame virtual characters are perceived as similar or different to their actual identity outside the game and to their idea of how they would like to be.

Other factors may affect players' identity exploration by means of their virtual selves. Therefore, other instruments will be included to measure participants' psychological distress, as well as more specific ones such as those targeting the level of immersion during the game and the main motivations that draw them to play.

As mentioned before, there are no empirical data regarding this issue yet. However, from a theoretical perspective, there can be several configurations of the relationships between actual, ideal, and virtual selves, leading to four types of online videogame players' virtual-self construal. The researchers have labeled each type of player according to how they would construe their virtual-self in relation to their actual and ideal selves.

* The first is the projection-type players, referring to those who construe their virtual identities as close to their ideal self, presumably to experiment with those attributes they perceive as more desirable. People who see themselves as more distant from their ideal selves could tend to fall under this category. This could serve as a strategy to obtain validation in the virtual environment while in the real world they mostly experience invalidation because their self is far from being ideal.
* The second type, named by the researchers as the exploration-type player. In contrast to the previous type, these players create virtual avatars that are more distant to both their actual and ideal selves as a way to explore alternative identities, not necessarily tied to their need to experience their ideal attributes, but rather for the enjoyment of exploring a completely different identity. Those players who already perceive themselves as very close to their ideal selves would be more likely to fall into this type since they would not feel such a need to experience their ideal self through a virtual character.
* For the third type, the term proximal-type player was chosen. It encompasses players whose virtual self resembles their actual self, regardless of its distance from the ideal self. A way this type of players may be encountered can be either when the level of immersion during the game experienced was too low for them to feel identified with their virtual avatar, or in the case, they played the game in a more competitive manner rather than as an interaction modality with other characters. Another explanation for why this type of player may not express a different aspect of their self through their virtual avatar may be because of a low interpersonal construct differentiation, which would make it harder for them to hold different instances of their identity.
* Lastly, there is the unspecified-type player, including those players whose virtual self is perceived as nearly equidistant from their actual and ideal selves without those two being necessarily close. Although mathematically, this may be a possible outcome from the actual-ideal-virtual self relationships, there is no theoretical premise that would account for this eventuality. Hence, it should be considered as a rare possibility to be carefully studied in case its prevalence was significant.

OBJECTIVES:

With this project, the researchers aim to explore how different identities may be explored thanks to virtual environments and how different factors may affect this identity exploration. More specifically, they want to assess how different people may create their virtual self differently and how these differences may be reflected in the previously predicted typology of players.

With regard to the player experience during the game, the researchers want to investigate whether the level of perceived immersion may influence a players' construal of their virtual self. Also, players' motivation for playing online videogames can lead to different experiences of the virtual self, and thus they want to investigate whether players' competitive orientation will influence the tendency to explore alternative identities through their virtual avatars as compared to those who enjoy more the social aspects. On the other hand, the researchers want to explore players' psychological distress and self-esteem as factors influencing the way they project their ideal self on their characters.

Another objective is to explore the role of cognitive conflicts or dilemmas in the participants' way of representing their self virtually. The researchers expect that a greater amount of internal conflict could influence the way players explore different identities through a virtual avatar since cognitive conflict can be a source of dissonance when a person construes their ideal self.

Secondarily, the researchers aim to study the role played by other variables on the way these players conceive their virtual self, such as their interpersonal construct differentiation, an indicator of cognitive complexity. However, this objective will be studied in a more exploratory manner, since there is still no theoretical background on the matter.

PROCEDURE

Participants will be contacted by making an online call on Internet forums, asking players who may be interested in participating to access an online survey using Qualtrics.

The survey will begin with the informed consent form, previously approved by the ethical committee. After reading and accepting the informed consent, participants will be presented with demographical and playing habits questions such as age, gender, country, employment status, average hours of play per week, whether or not they play professionally, and whether or not they have a record of severe mental illness or substance misuse. After that, they will answer the PENS, CORE-OM, and RSES questionnaires. The total duration of the survey will be 12 minutes, approximately.

After completing the survey, participants will be asked to indicate a date and hour when they will be available to appoint a virtual meeting conducted by Discord, one of the most widespread videoconference software within the gaming community. During this meeting, a predoctoral researcher will administrate the RGT to the participant, which will last for between 45 and 90 minutes. Each grid will be analyzed with the GRIDCOR 6.0 software, or with a more advanced version.

Participants will receive no payment for their collaboration, but upon completion of this project, those who wish it will receive a brief feedback report of their ratings.

For the analysis of the gathered data, the RStudio software will be used. The researchers will carry out a K-means cluster analysis in which they will specify participants to be clustered in three groups using their self-virtual and virtual-ideal discrepancies as the clustering criteria. Once the analysis has rendered the three clusters, the researchers will label them according to the previously mentioned player typologies. It is expected that there will be one group where the self-virtual discrepancy will be lower, indicating a proximal type of players. The researchers also expect that the two remaining clusters will be differentiated in terms of virtual-ideal discrepancy. Those with a higher discrepancy will be labeled as exploration-type and those with a lower discrepancy will be labeled as projection-type. Projection-type participants are also expected to have lower self-esteem than the other clusters.

A one-way ANOVA will be conducted to assess if there is a significant difference in self-virtual discrepancy between proximal-type players and the other two groups. Another one-way ANOVA will be carried out to assess check if there is a statistically significant difference between projection-type and exploration-type players in terms of self-ideal discrepancy. Through these analyses, the researchers expect to validate the typology of online videogame players based on their construal of their virtual-self.

After that, the researchers will carry out a multiple linear regression model, taking the self-virtual discrepancy as the outcome and using as independent variables the experienced immersion, taken from the correspondent scale from the PENS and the degree of cognitive complexity, inferred by means of the cognitive differentiation measure from the grid.

Another one-way ANOVA will be conducted to test whether if there are differences between the three groups in terms of their motivation toward the social or competitive aspects of the game, which will be inferred through the "relatedness" and "competence" scales from the PENS.

Finally, the researchers will carry out a multiple linear regression model within each group of players, taking the virtual-ideal discrepancy as the outcome for the projection and exploration types, whereas the outcome for the proximal type will be the self-virtual discrepancy, and using as predictors the level of cognitive conflict, the level of cognitive differentiation, and the measures of self-esteem, psychological distress, immersion, relatedness, and competence.

ELIGIBILITY:
Inclusion Criteria:

* Have an active World of Warcraft account.

Exclusion Criteria:

* Play World of Warcraft or any other game professionally
* Consume drugs while playing
* Previous or current record of severe mental disorders
* Any condition that renders a person unable to answer online or face-to-face surveys,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who play on a regular basis an online videogame that allows the creation of a customizable character. For this study, we are focusing on players of the game "World of Warcraft". We are focusing on general population from around the world who will be contacted online.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Repertory Grid: Self-Ideal Discrepancy | 1 week after Day 1
  Measured with the Repertory Grid Technique: It measures the distance between a person's ideal and actual self. A lower discrepancy indicates a greater self-esteem.
Repertory Grid: Self-Virtual Discrepancy | 1 week after Day 1
  Measured with the Repertory Grid Technique:The distance between the actual self and the virtual self. A lower discrepancy indicates a person's greater identification with their videogame character.
Repertory Grid: Virtual-Ideal Discrepancy | 1 week after Day 1
  Measured with the Repertory Grid Technique: The distance between the ideal self and virtual self. A lower discrepancy indicates a person's greater idealisation of their videogame character.

SECONDARY OUTCOMES:
Repertory Grid: Presence of implicative dilemmas | 1 week after Day 1
  Measured with the Repertory Grid Technique: Implicative dilemmas reflect conflictive relationships between a person's constructs that keep them from changing undesired traits or behaviors that they perceive as being closely linked to other desirable ones.
Repertory Grid: Presence of dilemmatic constructs | 1 week after Day 1
  Measured with the Repertory Grid Technique: Dilemmatic constructs can reflect a person's difficulty to discern how they would like to be in regard to the particular characteristic.
Repertory Grid: Interpersonal cognitive differentiation | 1 week after Day 1
  Measured with the Repertory Grid Technique: It is a measure of the complexity with which individuals construe their experiences, the degree they use nuances (or not) in discriminating among self and others.
PENS: Immersion | Day 1.
  Measured with the Player Experience of Need Satisfaction questionnaire: It indicates the level of immersion experienced by a person when they play a specific videogame. The score can range from 9 to 63.
PENS: Relatedness | Day 1.
  Measured with the Player Experience of Need Satisfaction questionnaire: It indicates how much a specific videogame fulfills a person's necessity for social interaction. The score can range from 3 to 21.
PENS: Competence | Day 1.
  Measured with the Player Experience of Need Satisfaction questionnaire: It indicates how much a specific videogame fulfills a person's necessity for competitivity and achievement. The score can range from 3 to 21.
Psychological Distress | Day 1.
  Measured with the Clinical Outcomes in Routine Evaluation - Outcome Measure questionnaire: It indicates a person's levels of psychological well-being experienced on different dimensions. The total score can range from 0 to 136, and the mean score ranges from 0 to 4.
Self-esteem | Day 1.
  Measured with the Rosenberg self-esteem scale: It can range from 10 to 40 and it is an indicator of a person's level of self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas Viaplana, Study Director — University of Barcelona
Locations (1):
- University of Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bessiere K, Seay AF, Kiesler S. The ideal elf: identity exploration in World of Warcraft. Cyberpsychol Behav. 2007 Aug;10(4):530-5. doi: 10.1089/cpb.2007.9994. PMID 17711361
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Feixas, G., Bach, L., & Laso, E. (2004). Factors affecting interpersonal construct differentiation when measured using the repertory grid.Journal of Construc- tivist Psychology,17, 297-311.
- [Background] Feixas, G. & Cornejo, J.M. (1996). Manual de la técnica de rejilla mediante el programa RECORD ver. 2.0 (2a ed.) Barcelona: Paidós.
- [Background] Fransella, F., Bell, R. & Bannister, D. (2004). A manual for repertory grid technique (2nd edition). Chichester: Wiley.
- [Background] Garcia-Gutierrez, A. & Feixas, G. (2018). GRIDCOR: A Repertory Grid Analysis Tool (Version 6.0) [Web application]. Retrieved from http://www.repertorygrid.net/en
- [Background] Gilbert, R., Thadani, V., Handy, C., Andrews, H., Sguigna, T., Sasso, A. & Payne, S. (2014). The psychological functions of avatars and alt(s): A qualitative study. Computers in Human Behavior, 32, pp. 1-8.
- [Background] Hu, C., Zhao, L. & Huang, J. (2015). Achieving self-congruency? Examining why individuals reconstruct their virtual identity in communities of interest established within social network platforms. Computers in Human Behavior, 50, pp. 465-475.
- [Background] Johnson, D., Gardner, M. J. & Perry, R. (2018). Validation of two game experience scales: The Player Experience of Need Satisfaction (PENS) and Game Experience Questionnaire (GEQ). International Journal of Human-Computer Studies, 118, pp.38-46.
- [Background] Kovářová, M., & Filip, M. (2015). Integrating the differentiated: A review of the personal construct approach to cognitive complexity. Journal of Constructivist Psychology, 28(4), 342-366.
- [Background] Montesano A, Lopez-Gonzalez MA, Saul LA, Feixas G. A review of cognitive conflicts research: a meta-analytic study of prevalence and relation to symptoms. Neuropsychiatr Dis Treat. 2015 Dec 4;11:2997-3006. doi: 10.2147/NDT.S91861. eCollection 2015. PMID 26675503
- [Background] Przybylski AK, Weinstein N, Murayama K, Lynch MF, Ryan RM. The ideal self at play: the appeal of video games that let you be all you can be. Psychol Sci. 2012 Jan 1;23(1):69-76. doi: 10.1177/0956797611418676. Epub 2011 Dec 14. PMID 22173739
- [Background] Ribeiro, J. C. (2009). The increase of the experiences of the self through the practice of multiple virtual identities. PsychNology Journal, 7 (3), pp. 291-302.
- [Background] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton: Princeton University Press.
- [Background] Stevens MJ. Prescott Lecky: pioneer in consistency theory and cognitive therapy. J Clin Psychol. 1992 Nov;48(6):807-11. doi: 10.1002/1097-4679(199211)48:63.0.co;2-c. PMID 1452769
- [Background] Walker BM, Winter DA. The elaboration of personal construct psychology. Annu Rev Psychol. 2007;58:453-77. doi: 10.1146/annurev.psych.58.110405.085535. PMID 16903803
- See also: Research Group Conducting the Study — http://www.ub.edu/ipcs/en/